CLINICAL TRIAL: NCT04097314
Title: A Randomised, Double-blind, Placebo-controlled, Cross-over Trial of Zibotentan in Microvascular Angina
Brief Title: Precision Medicine With Zibotentan in Microvascular Angina
Acronym: PRIZE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); King's College London (Other); University of Oxford (Other); Oxford University Hospitals NHS Trust (Other); University of Cambridge (Other); Papworth Hospital NHS Foundation Trust (Other Government); Blackpool Teaching Hospitals NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); AstraZeneca (Industry); Siemens Healthcare Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GN18CA068
Record Dates: First submitted 2019-07-05; First posted 2019-09-20 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-04

CONDITIONS: Microvascular Angina
Keywords: Microvascular Angina; Angina; Endothelin; MVA; Impaired Exercise Intolerance
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris | interventions — ZD4054

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zibotentan (Experimental)
  Interventions: Drug: Zibotentan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Zibotentan — 10mg OD Zibotentan
  Arms: Zibotentan
Drug: Placebo oral tablet — Placebo
  Arms: Placebo

SUMMARY:
Microvascular angina (MVA) is caused by abnormalities of the small vessels in the heart. Endothelin is a small chemical that circulates and accumulates in the blood vessel walls, causing them to narrow or go into spasm and thicken in the longer term especially as levels of endothelin increase. As a result, patients experience pain, psychological burden and an inability to carry out daily activities.

Originally developed by AstraZeneca for cancer treatment, prior research has confirmed that Zibotentan relaxes the small blood vessels of patients with MVA which lends support to the idea that Zibotentan may bring some benefits to patients with MVA. This trial therefore proposes to look into re-purposing zibotentan as a new treatment for patients with MVA. The primary objective is to assess the effect of add-on treatment with Zibotentan to treadmill exercise times in adult patients with MVA and impaired exercise intolerance. Zibotentan could provide a new treatment pathway for patients, as well as be made available to the NHS at substantially lower cost than the currently used medications.

The trial aims to initially invite approx. 356 participants for genetic testing. A minimum of 100 participants will go forward into the main study, receiving either 10mg zibotentan or a dummy matched tablet (placebo) daily over two 12 weeks periods of each, completing their final visit at week 34. The study assessments will involve a health check at each visit, including information on the patient's wellbeing, blood tests, some quality of life questionnaires, and an exercise test. Participants will also have the option to consent to additional sub-study cardiovascular MRI scanning. Finally, participants will be invited to provide consent for long-term follow-up (maximum 20 years) of their electronic medical records (no additional patient contact).

DETAILED DESCRIPTION:
The study design publication is available at https://pubmed.ncbi.nlm.nih.gov/32942043/

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Microvascular angina - as defined by COVADIS diagnostic criteria for microvascular angina.
3. Able to comply with study procedures.
4. Written informed consent.

Exclusion Criteria:

1. Exercise tolerance >540 seconds in men and >430 seconds in women (i.e. actual exercise duration (s) achieved on the Bruce protocol commensurate with predicted), or, lack of anginal symptoms and/or ST-segment depression (0.1 mV) limiting exercise.
2. Non-cardiovascular exercise-limiting problem e.g. morbid (or severe) obesity (BMI ≥40.0 kg/m2)
3. Genotype not available
4. Women who are pregnant, breast-feeding or of child-bearing potential (WoCBP) without a negative pregnancy test and who are unwilling or unable to follow the reproductive restrictions and use highly effective contraception as defined in Appendix 3 of the protocol for the duration of the study treatment and 30 days after last dose of study drug.
5. Men who are sexually active with a WoCBP who are unwilling to use condoms or other highly effective methods of contraception for the duration of study treatment and for 14 weeks after last dose of study drug.
6. Heart failure (New York Heart Association Grade ≥II i.e. mild symptoms and slight limitation during ordinary activity)
7. Recent (<3 months) myocardial infarction
8. A history of epilepsy, other CNS adverse events, neurologic symptoms or signs consistent with spinal cord compression or CNS metastases.
9. Moderate or more severe renal impairment (GFR < 45 mL/min)
10. Liver disease with a Child-Pugh score of A (5-6 points) or higher
11. Participation in another intervention study involving a drug within the past 90 days or 5 half-lives whichever is longer (co-enrolment in observational studies is permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
EFFICACY - Exercise Testing (treadmill exercise time, seconds) | 34 weeks
  The primary outcome is the treadmill exercise time (TET) measured in seconds using the Full Bruce protocol, a measure of aerobic capacity that reflects disease severity. A within-subject improvement in exercise time (tested at week 10 (baseline), week 22 (crossover) and week 34 (final visit)) of 30 seconds is considered clinically relevant.

SECONDARY OUTCOMES:
EFFICACY - Health Status QLQ (Seattle Angina Questionnaire) | 34 weeks
  Seattle Angina Questionnaire (SAQ) Summary Score and component scores (Angina Limitation, Angina Stability, Angina Frequency, Treatment Satisfaction and Quality of Life) will be recorded at all study visits.
EFFICACY - Health Status QLQ (Illness Perception - Brief IPQ) | 34 weeks
  Brief Illness Perception Questionnaire (Brief IPQ), a nine-item scale designed to rapidly assess the cognitive and emotional representations of illness taken at all study visits.
EFFICACY - Health Status QLQ (Anxiety/depression - PHQ4) | 34 weeks
  The Four-Item Patient Health Questionnaire (PHQ-4) for Anxiety and Depression is a validated tool for detecting both anxiety and depressive disorders and will administered at all study visits
EFFICACY - Health Status QLQ (Treatment satisfaction - TSQM) | 34 weeks
  The 14-item Treatment Satisfaction Questionnaire for Medication (TSQM) is a reliable and valid instrument to assess patients' satisfaction with medication, providing scores on four scales - side effects, effectiveness, convenience and global satisfaction and will administered at all study visits
EFFICACY - Health Status QLQ (EQ5D-5L) | 34 weeks
  The 5-item EuroQol Group EQ5D-5L is a validated questionnaire comprising mobility, self-care, usual activities, pain/discomfort and anxiety/depression to quantitatively assess patient's self-reported health status and will be administered at each study visit.
FEASIBILITY - Withdrawal Rate | 34 weeks
  Participant withdrawal rate from study will be measured throughout.
SAFETY - SAEs | 34 weeks
  Number of Participants With Treatment-Related Adverse Events as Assessed and reported by local study teams throughout trial.
EFFICACY - Exercise Testing (time,sec to 1mm ST-depression) | 34 weeks
  Within-subject improvements in time (seconds) to 1 mm ST-depression during exercise tolerance testing will be assessed using the Full Bruce protocol. Assessments will be during screening, week 10 (baseline), week 22 (crossover) and week 34 (final visit).
EFFICACY - Exercise Testing (maximum ST-segment deviation, mV) | 34 weeks
  Within-subject improvements in maximum ST-segment deviation (mV) during exercise tolerance testing will be assessed using the Full Bruce protocol. Assessments will be during screening, week 10 (baseline), week 22 (crossover) and week 34 (final visit).
EFFICACY - Exercise Testing (Time (s) to 75% of max age-related heart rate during exercise) | 34 weeks
  Within-subject improvements in time (seconds) to 75% of max age-related heart rate during exercise tolerance testing will be assessed using the Full Bruce protocol. Assessments will be during screening, week 10 (baseline), week 22 (crossover) and week 34 (final visit).
EFFICACY - Exercise Testing (Metabolic equivalent (METs) | 34 weeks
  Within-subject improvements in metabolic equivalent (METs) during exercise tolerance testing will be assessed using the Full Bruce protocol. Assessments will be during screening, week 10 (baseline), week 22 (crossover) and week 34 (final visit). The resting metabolic rate is defined as 3.5 ml O2/kg/min (METs).
EFFICACY - Exercise Testing (DUKE Score) | 34 weeks
  Within-subject improvements in Duke treadmill score (DTS) during exercise tolerance testing will be assessed using the Full Bruce protocol. Assessments will be during screening, week 10 (baseline), week 22 (crossover) and week 34 (final visit). Duke treadmill score is defined as maximum exercise time in minutes - (5 × the maximal net ST-segment deviation in mm during or after exercise) - (4 × the treadmill angina index (where 0 = no angina, 1 = non-limiting angina, 2 = exercise limiting angina).

OTHER OUTCOMES:
EFFICACY - Pharmacodynamics (Exploratory) | 34 weeks
  Blood samples will be obtained at weeks 10, 22 and 34 to measure circulating concentrations of mechanistic biomarkers. These analyses are intended to provide insights into the mechanisms of treatment-related efficacy and safety responses.These measurements will be considered an exploratory endpoint.
EFFICACY - Pharmacokinetics (Exploratory) | 34 weeks
  Blood samples will be obtained at weeks 10, 22 and 34 to measure steady-state plasma concentrations of zibotentan with a validated assay. These measurements will be considered an exploratory endpoint.
EFFICACY - Angina Diary (Exploratory) | 34 weeks
  A novel, bespoke questionnaire for the diagnostic classification of patients with ischaemia with non-obstructive coronary artery disease (INOCA) and their treatment response will be assessed as an exploratory outcome. Patients are asked to complete this diary every time they suffer angina symptoms over the course of the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morrow A, Young R, Abraham GR, Hoole S, Greenwood JP, Arnold JR, El Shibly M, Shanmuganathan M, Ferreira V, Rakhit R, Galasko G, Sinha A, Perera D, Al-Lamee R, Spyridopoulos I, Kotecha A, Clesham G, Ford TJ, Davenport A, Padmanabhan S, Jolly L, Kellman P, Kaski JC, Weir RA, Sattar N, Kennedy J, Macfarlane PW, Welsh P, McConnachie A, Berry C; PRIZE Study Group. Zibotentan in Microvascular Angina: A Randomized, Placebo-Controlled, Crossover Trial. Circulation. 2024 Nov 19;150(21):1671-1683. doi: 10.1161/CIRCULATIONAHA.124.069901. Epub 2024 Sep 1. PMID 39217504